CLINICAL TRIAL: NCT02502955
Title: Virtual Autopsy in Cardiology, Cardio- and Vascular-Surgery
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: VA-4 Cardio
Record Dates: First submitted 2015-06-16; First posted 2015-07-20 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Death
Keywords: Quality Control; Cardiosurgery; Cardiology; Vascular Surgery; ICU
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Comparison autopsy methods — Comparison of post-mortem angiography/virtual autopsy and medical autopsy

SUMMARY:
Today complex vascular and cardiological interventions are performed in severely ill patients.

Autopsy is the reference standard for quality control for almost two centuries, but autopsy rates for patients dying in hospitals are decreasing rapidly.

Virtual autopsy has shown to be a good alternative for classic autopsy.

DETAILED DESCRIPTION:
Patients dying within 96h after a cardiological intervention of a cardio-/vascular-surgery are eligible to be included in the study.

If the next of kin give oral informed consent a virtual autopsy based on a CT angiography followed by a classic medical autopsy will be performed.

Ante mortem findings will be compared to findings from both autopsy methods and presented to the clinicians.

Primary outcome will be the inter-method agreement. Secondary outcome will be the satisfaction of the clinicians evaluated by a standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older AND
* dying after a cardiological intervention or a cardio-/vascular surgery AND
* oral informed consent from next of kind

Exclusion Criteria:

* not fulfilling all inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients dying after a cardiological intervention or a cardio-/vascular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Agreement of virtual autopsy and medical autopsy (inter-method agreement) | 1 week
  Diagnoses made by virtual autopsy will be compared to diagnoses made by classic autopsy.

SECONDARY OUTCOMES:
Quality evaluation (satisfaction of the clinicians evaluated by a standardized questionnaire) | 2 weeks
  Diagnoses made by any autopsy method will be compared to ante mortem diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Wichmann, MD, Principal Investigator — Department of Intensive Care Medicine, University Medical Center Hamburg
Locations (1):
- Department of Intensive Care Medicine, University Medical Center Hamburg-Eppendorf (UKE), Hamburg, Germany